CLINICAL TRIAL: NCT03481413
Title: Patient Specific Optimized Therapy Post-Market Clinical Follow-up Study
Acronym: PSOT-PMCF
Status: Terminated | Type: Observational
Why Stopped: Philips decided to wind down the EPD Solutions business
Sponsor: EPD Solutions, A Philips Company (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-KODEX-0007; NCT03619018 (obsolete NCT alias)
Record Dates: First submitted 2018-03-05; First posted 2018-03-29 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Arrythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Ablation — Ablation therapy for cardiac arrhythmias

SUMMARY:
Study to evaluate the safety and procedural performance of the KODEX - EPD System when used in the treatment of cardiac arrhythmias. An additional objective is to develop patient specific optimized therapy (PSOT PMCF) via machine learning to improve future treatment of cardiac arrhythmias (PSOT).

DETAILED DESCRIPTION:
PSOT PMCF is a prospective, multi-center, non-randomized, open label, single arm observational/ registry clinical study. Consented subjects who are scheduled to undergo an ablation procedure due to an arrhythmia will be enrolled in the clinical study. The clinical study consists of a standard-of-care index ablation procedure and following up subjects for 12 months to evaluate product safety. The index ablation procedure will be performed using the KODEX - EPD System in conjunction with compatible therapeutic and diagnostic catheters. Electrophysiologists should follow current, local, and expert consensus guidelines when treating subjects.

The PSOT Sub-Study Secondary System is a sub-study of the PSOT PMCF study. The objective of the sub-study is to collect data for the evaluation of the performance of new software features via a secondary system in subjects undergoing standard of care catheter-based endocardial mapping for cardiac arrhythmia's using a commercial KODEX EPD Mapping System.

The KODEX-EPD system in this clinical investigation will have a Primary/Secondary configuration. Data collection and processing will be done on the Primary system in the interventional lab with market released software and the Primary system will be used to guide therapy. Data from the Primary system will be transferred to a second (Secondary) workstation in the control/observation room via unidirectional communication and data on the Secondary system will be processed with non-released software.

Results from this sub-study will be used to support the development and refinement of new software features. It is not the purpose of this sub-study to obtain CE mark.

The primary endpoint of the sub-study is data collection of the KODEX-EPD non-released features from a secondary system.

ELIGIBILITY:
Inclusion Criteria:

1. . Subjects who are eligible for an ablation procedure based on local guidelines,
2. . Subjects must be 18 years of age or above and at a legal age to give informed consent specific to state and national laws
3. . Subjects must be able and willing to comply with all follow-up requirements

Exclusion Criteria

1. . Women who are pregnant (as evidenced by pregnancy test if pre-menopausal; method of assessment upon the discretion of the investigator),
2. . Life expectancy less than 12 months,
3. . Participation in a concurrent clinical study without prior approval from EPD Solutions.
4. . Any contra-indication to use KODEX-EPD System per User Manual.
5. . Unrecovered/unresolved adverse events from any previous invasive procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Arrhythmia patients indicated for EP procedures.
  Both male and female subjects who meet all eligibility criteria and give written informed consent will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 566 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Acute safety event rate when using the KODEX - EPD System | 7 days
  The primary safety event rate will be measured against a pre-specified performance goal of 12% and include serious system- or procedure-related adverse events occurring within 7 days of the index procedure
The success rate of the index ablation procedure. | Index procedure
  A procedure is defined as successful if the following conditions are met:
  1. KODEX - EPD System was the only mapping system used in the index ablation procedure.
  2. The primary arrhythmia was terminated and validated by operators' standard clinical practice (e.g., pacing).

SECONDARY OUTCOMES:
12-month safety event rate when the KODEX - EPD System was used in the index ablation procedure and any additional unplanned follow-up procedures. | 12 months
  The primary safety event-free rate will be measured against a pre-specified performance goal of 15% and include serious system- or procedure-related adverse events occurring within 12 months from the initial index procedure.
Develop PSOT for cardiac arrhythmia patients. | Index procedure
  PSOT PMCF will find appropriate functions to map predictor variables (e.g., subject demographics, arrhythmia type, ablation energy source, etc.) to target variables (e.g., procedure success, adverse events, etc.) with the goal of improving efficacy and minimizing adverse events for future cardiac arrythmia subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Anish Amin, MD, Principal Investigator — OhioHealth Riverside Methodist Hospital; Yitschak Biton, MD, Principal Investigator — Hadassah Medical Organization; Min Tang, MD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (22):
- United States (6):
  - Dignity Health Research Institute, Sacramento, California
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - NYU Langone Health, New York, New York
  - OhioHealth Riverside Methodist Hospital, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
- Belgium (2):
  - Onze Lieve Vrouw Ziekenhuis Aalst, Aalst
  - AZ Sint Jan, Bruges
- Germany (5):
  - Herz- und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen
  - HELIOS Klinikum Erfurt, Erfurt
  - Klinikum Fürth, Fürth
  - Universitätsklinikum Hamburg-Eppendorf (UKE Hamburg), Hamburg
  - Kardiologische Gemeinschaftspraxis am Park Sanssouci, Potsdam
- Israel (2):
  - Hadassah University Medical centrum, Jerusalem
  - Shaare Zedek Medical Center, Jerusalem
- Italy (2):
  - Clinica Montevergine, Mercogliano
  - Monzino Cardiologic Centre, University of Milan., Milan
- Netherlands (3):
  - Catharina Ziekenhuis, Eindhoven
  - Maastricht UMC, Maastricht
  - Sint Anthonius ziekenhuis, Utrecht
- Fondazione Cardiocentro Ticino, Lugano, Switzerland
- Glenfield Hospital-University of Leicester, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No